CLINICAL TRIAL: NCT04939298
Title: Ultrasound Evaluation of Abdominal Muscle Thickness During Mechanical Ventilation
Acronym: ABDO-VM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Roanne (Other)
Collaborators: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020/01; 2020-A03186-33 (Other: ANSM)
Record Dates: First submitted 2021-06-11; First posted 2021-06-25 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Ventilation Therapy; Complications
Keywords: abdominal muscles; ultrasound
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients under mechanical ventilation (Experimental): Ultrasound evaluation of the variation of thickness of abdominal muscles after 7 days of mechanical ventilation
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Ultrasound evaluation of the variation of thickness of abdominal muscles after 7 days of mechanical ventilation.

SUMMARY:
Weakness of respiratory muscles is frequent after several days of mechanical ventilation. Thereby an acquired diaphragm weakness has been demonstrated, linked to an atrophy which may be identified by a decrease of muscle thickness in echography. This study aims to evaluate with ultrasound the variation of thickness of abdominal muscles after 7 days of mechanical ventilation.

DETAILED DESCRIPTION:
Weakness of respiratory muscles is frequent after several days of mechanical ventilation. Thereby an acquired diaphragm weakness has been demonstrated, linked to an atrophy which may be identified by a decrease of muscle thickness in echography. Weakness of expiratory muscles is also frequent after 7 days of mechanical ventilation, however his cause is not clear: is it present at admission notably in elderly patients, or acquired on mechanical ventilation ? Ultrasound allows to measure the thickness of abdominal muscles which correlates with their strength. This study aims to evaluate with ultrasound the variation of thickness of abdominal muscles after 7 days of mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Patient affiliated or entitled to a social security plan
* Expected duration of mechanical ventilation > 7 days
* Trusted person/relative who has signed a consent to participate in the study

Exclusion Criteria:

* Patient with a pre-existing neuromuscular pathology
* No access to ultrasound Windows (dressing, drainages...)
* Patient transferred from another intensive care unit
* Patient Under guardianship or curators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2023-11-16 (Actual)

PRIMARY OUTCOMES:
Thickness of the abdominal muscles (mm) | Day 7
  It is the sum of the thickness of rectus abdominal muscle + external oblique + internal oblique + transverse muscles.

SECONDARY OUTCOMES:
Thickness of the rectus abdominal muscles (mm) | Day 7
  Thickness of the rectus abdominal muscles (mm) by ultrasound measurement.
Thickness of the external oblique abdominal muscles (mm) | Day 7
  Thickness of the external oblique abdominal muscles (mm) by ultrasound measurement
Thickness of the internal oblique abdominal muscles (mm) | Day 7
  Thickness of the internal oblique abdominal muscles (mm) by ultrasound measurement
Thickness of the transverse abdominal muscles (mm) | Day 7
  Thickness of the transverse abdominal muscles (mm) by ultrasound measurement
Diaphragmatic thickness (mm) | Day 7
  Diaphragmatic thickness (mm) measured by ultrasound
Diaphragmatic thickness (mm) | Immediately after the successful extubation of the patient
  Diaphragmatic thickness (mm) measured by ultrasound
Number of day with a contraction of the transverse abdominal muscle | From day 1 to day 7
  Ultrasound search for a contraction of the transverse abdominal muscle during the morning clinical examination each day from D1 to D7
Caught peak expiratory flow (CPEF) (cmH2O) | Day 7
  Only for conscious patients, responding to the simple command and tolerating minimal respiratory support (inspiratory support 7 cmH20, Pep 0 cmH20) caught peak expiratory flow (CPEF) measurement
Maximum expiratory pressure (l/min) | Day 7
  Only for conscious patients, responding to the simple command and tolerating minimal respiratory support maximum expiratory pressure (PE max) measurement
Thickness of the external oblique abdominal muscle (mm) | Immediately after the successful extubation of the patient
  External oblique abdominal muscle by ultrasound measurement
Thickness of the internal oblique abdominal muscle (mm) | Immediately after the successful extubation of the patient
  Internal oblique abdominal muscle by ultrasound measurement
Thickness of the transverse abdominal muscle (mm) | Immediately after the successful extubation of the patient
  Transverse abdominal muscle by ultrasound measurement
Thickness of the rectus abdominal muscle (mm) | Immediately after the successful extubation of the patient
  Rectus abdominal muscle by ultrasound measurement
Number of day between day 7 and successful extubation day (days) | From Day 7 to the day when the patient will be extubated successfully
Duration of sedation (Day) | At intensive care unit discharge
Duration of curarization (Day) | At intensive care unit discharge

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Beuret, MD, Principal Investigator — HOPITAL DE ROANNE
Locations (1):
- Centre Hospitalier de Roanne, Roanne, France

IPD SHARING:
Plan to Share IPD: No